CLINICAL TRIAL: NCT00792077
Title: A Pilot Open Label Study to Investigate the Effect of Cytotoxic Therapy and/or Radiotherapy Including Lenalidomide on Cancer Related Sleep Disturbances in Chronic Lymphocytic Leukemia (CLL) and Breast Cancer Patients Experiencing Clinically Significant Fatigue
Brief Title: A Pilot Study to Investigate the Effect of Cytotoxic Therapy and/or Radiotherapy on Cancer Related Sleep Disturbances in CLL and Breast Cancer Patients Experiencing Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0945; NCI-2012-01661 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Leukemia; CLL
Keywords: Leukemia; Lenalidomide; Actigraph; Sleep Test Study; Chronic Lymphocytic Leukemia; CC-5013; Revlimid
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sleep time (Experimental): Assessment of patients with chronic lymphocytic leukemia (CLL) experience severe cancer related fatigue (CRF):
  Lenalidomide + Actigraph + Questionnaire + Sleep Test
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 5 mg daily for 56 days.
  Other Names: CC-5013; Revlimid

SUMMARY:
The goal of this clinical research study is to learn if treatments to kill cancer cells including lenalidomide and/or radiation therapy can help to control symptoms such as sleep problems and fatigue in patients with chronic lymphocytic leukemia (CLL) and/or breast cancer.

DETAILED DESCRIPTION:
In this study, researchers are trying to learn if treatments to kill cancer cells such as lenalidomide and/or radiation therapy can also help to control sleep problems and fatigue in patients with CLL and/or breast cancer.

Study Procedures:

If you are found to be eligible to take part in this study, before you begin taking chemotherapy on Day 1, the following tests and procedures will be performed:

* Blood (about 2 tablespoons) will be drawn to learn about the relationship between changes in specific protein levels in the blood, your level of fatigue, and sleep problems.
* Your complete medical history will be recorded.
* You will have a physical exam.
* You will also complete 4 questionnaires that will ask you questions about your symptoms and your sleep patterns. They will take 20-30 minutes to complete in total.

From Day 1 through the end of 1st cycle (+/- 3 days), you will wear a watch that records your body movements. This is called an actigraph.

On Day 15 (+/- 3 days), you will be called by a member of the research staff. During these calls, you will complete the 4 questionnaires that ask about symptoms you are having and about your sleep patterns.

On Day 29 (+/- 3 days) and end of 1st cycle (+/- 3 days), you will have a clinic visit. At this visit, you will complete the 4 questionnaires that ask about symptoms you are having and your sleep patterns. Blood (about 2 tablespoons) will also be drawn to learn about the relationship between changes in protein levels in the blood, your level of fatigue, and sleep problems.

Sleep Tests:

You will have a sleep test before starting chemotherapy on Day 1 and again on end of 1st cycle (+/- 3 days). The sleep test is done overnight in a sleep lab.

A sleep study, called a polysomnogram, is a test that records a person's physical state during various stages of sleep and wakefulness. The study provides information about a person's sleep stages, body position, blood oxygen levels, breathing events, muscle tone, heart rate, snoring, and general sleep behavior.

When you arrive at the Sleep Center Laboratory you will be shown to your private room. You will complete a questionnaire that will ask questions about how much you slept the night before, how active you have been, and about any caffeine or alcohol you may have had. The questionnaire will take about 5 minutes to complete.

The member of the sleep lab staff will connect sensors that will record your brain waves, muscle tone, eye movements, air flow, and limb movements while you sleep. The sensors are applied to specific areas of your body with paste and gauze or tape. The monitoring equipment is painless and should not interfere with your sleep.

It is not a problem to have a drink of water or to use the restroom during the sleep study. The member of the sleep lab staff will monitor the sleep study from another room throughout the night and will wake you in the morning to remove the sensors.

In the morning, you will complete a questionnaire about how you slept and how you are feeling. It will take about 5 minutes to complete.

Length of Study:

You will be on study up to end of 1st cycle (+/- 3 days).

This is an investigational study. Sleep studies are a standard test for patients with sleep problems.

The blood tests performed for this study and the sleep test will be performed at no cost to you.

Up to 12 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Describe fatigue as being present every day for most of day for a minimum of 2 weeks and rate fatigue greater than or equal to 4 on a 0-10 scale, in which 0= no fatigue and 10=worst possible fatigue as assessed by MD Anderson symptom Inventory(MDASI).
2. Have diagnoses of CLL and started on a new cytotoxic therapy or breast cancer receiving new cytotoxic or radiation therapy
3. Patients will be eligible to participate in this study if they rate sleep disturbance greater than or equal to 4 on a 0-10 scale, in which 0= disturbed sleep is not present and 10 = disturbed sleep as bad as you can imagine as assessed by MDASI.
4. Have a MDAS of 13 or less.
5. Able to understand the description of the study and give written informed consent.

Exclusion Criteria:

1. Patients who are unable to complete the assessment measures or refuse to participate
2. Patients with known history of brain metastasis.
3. Patients with known history of sleep apnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennurajalingam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Chronic lymphocytic leukemia were recruited from the Leukemia Clinic at the University of Texas MD Anderson Cancer Center.
Groups:
- Lenalidomide: Participants received lenalidomide 5mg orally daily for 57 +/- 3 days
Period: Overall Study
Arm/Group | Lenalidomide
Started | 6
Day 15+/- 3 Days | 6
Day 29+/-3 Days | 6
Day 43+/-3 Days | 6
Day 57+/-3 Days | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6
Marital Status [Count of Participants; unit: Participants]
  Divorced | 2
  Married | 3
  Separated | 1
Employment Status [Count of Participants; unit: Participants]
  Full Time | 2
  Medical Leave | 1
  Part time | 1
  Unemployed | 2

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time as Measured by Polysomnography (PSG)
Description: Polysomnography (PSG) was done to measure the total sleep time in minutes. It was measured as a change in total sleep time between the before and after 1st cycle of treatment with Lenalidomide.
Time Frame: before and after 1st cycle of Lenalidomide treatment, up to 8 weeks
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
Minutes | -25.5 [-46.0 to -15.0]

2. Secondary Outcome: The Functional Assessment of Chronic Illness Therapy-Fatigue Subscale Score
Description: The FACIT-F subscale is a validated measure of fatigue. In the FACIT-F, the patient rates the intensity of their fatigue and its related symptoms on a scale of 0 to 4. The total score can range between 0 and 52, with higher scores denoting less fatigue. The score 0= worst fatigue possible, 52 indicates no fatigue. The scores reported is the median (IQR) change at 8 weeks compared to baseline.
Time Frame: before and after 1st cycle of Lenalidomide treatment, up to 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
score on a scale | 4 [-11 to 8]

3. Secondary Outcome: Epwort Sleep Scale
Description: The Epworth sleep scale is an 8-item questionnaire designed to asses general level of daytime sleepiness, and scores on this instrument range form 0-24, with higher scores indicating greater sleepiness. It was measured as a change in total score between the before and after 1st cycle of treatment with Lenalidomide.
Time Frame: before and after 1st cycle of Lenalidomide treatment, up to 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
score on a scale | -1 [-3 to 1]

4. Secondary Outcome: ECOG Performance Status
Description: This criteria is used to assess how a patient's disease is progressing and to assess how the disease affects the daily living abilities of the patient. The scores on this instrument range from 0-5 (0=fully active and 5=dead), with higher scores indicating poorer performance. It was measured as a change in performance status between before and after 1st cycle of treatment with Lenalidomide.
Time Frame: before and after first cycle of Lenalidomide treatment, up to 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
score on a scale | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: before and after 1st cycle of Lenalidomide treatment, up to 8 weeks
Arm/Group | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-07-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT00792077/Prot_SAP_000.pdf